CLINICAL TRIAL: NCT06840704
Title: Immunonutrition in Reducing Acute Esophagitis After Thoracic Radiotherapy in Lung Cancer: a Prospective, Randomized, Controlled, Open-label Clinical Trial
Brief Title: Immunonutrition Reduces Acute Esophagitis After Thoracic Radiotherapy in Lung Cancer
Acronym: Relief
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, HuaiLiu, Prof., Hunan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT128
Record Dates: First submitted 2025-02-08; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer; esophagitis; immunonutrition; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Esophagitis | interventions — Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral immunonutrition (Experimental): Oral immunonutrition (Oral Impact®, Nestlé), 250 ml per bottle, with a dosage of 2 bottles per day, starting on the day of radiotherapy and continuing for three weeks after radiotherapy.
  Interventions: Dietary Supplement: Oral immunonutrition
- Standard nutrition (No Intervention): If the patient has concurrent nutritional risks, routine nutritional therapy (no immunonutrition) can be provided under the guidance of a nutritionist.

INTERVENTIONS:
Dietary Supplement: Oral immunonutrition — Oral immunonutrition (Oral Impact®, Nestlé), 250 ml per bottle, with a dosage of 2 bottles per day, starting on the day of radiotherapy and continuing for three weeks after radiotherapy.
  Arms: Oral immunonutrition

SUMMARY:
This study aims to evaluate the efficacy of immunonutrition in reducing acute esophagitis after thoracic radiotherapy in lung cancer.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, open-label clinical trial, which aimed to explore the efficacy and safety of oral immunonutrition therapy in reducing acute esophagitis after thoracic radiotherapy in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in this clinical study, understands the study procedures, and is able to provide written informed consent.
2. Age ≥ 18 years.
3. Pathologically confirmed diagnosis of lung cancer, including non-small cell lung cancer and small cell lung cancer.
4. Indication for thoracic radiotherapy, with the esophagus within 1 cm of the PTV.
5. Prescription dose for the PTV: 60-70 Gy once daily (2 Gy/Fx), 45 Gy twice daily (1.5 Gy/Fx, with intervals exceeding 6 hours), or 45 Gy once daily (3 Gy/Fx).
6. Ability to orally intake food normally.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
8. The volume of both lungs receiving more than 20 Gy (V20) should not exceed 30% of the total lung volume.
9. Expected survival of more than 3 months.
10. Laboratory test results during the screening period:

    Complete blood count: ANC ≥ 1.5 × 10^9/L; PLT ≥ 80 × 10^9/L; Hb ≥ 90 g/L. Blood biochemistry: TBIL ≤ 1.5 × ULN; ALT and AST ≤ 2 × ULN; BUN and Cr ≤ 1.5 × ULN, with creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula).
11. Female subjects of childbearing potential, male subjects, and partners of male subjects agree to use reliable contraceptive methods during the study period (such as abstinence, sterilization, oral contraceptives, or other contraceptive measures).

Exclusion Criteria:

1. Previous history of thoracic radiotherapy.
2. Suspected or confirmed tumor invasion of the esophagus.
3. Patients with other primary tumors.
4. History of esophageal cancer, gastric cancer, or prior esophageal surgery.
5. Concurrent active reflux esophagitis.
6. Current regular use of immunonutrition (e.g., Oral Impact®).
7. Patients with severe cardiovascular or cerebrovascular diseases, or comorbidities such as liver or kidney diseases.
8. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study period.
9. Concurrent active autoimmune diseases requiring treatment.
10. Known history of human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS).
11. Any medical (e.g., pulmonary, metabolic, endocrine, or neurological diseases, congenital disorders, etc.), psychiatric, or social condition that, in the investigator's judgment, may interfere with the subject's rights, safety, health, or ability to provide informed consent, cooperate and participate in the study, or interfere with the evaluation of the study drug, interpretation of patient safety, or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of grade 2 or higher acute esophagitis | 3 months
  Assessed according to National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

SECONDARY OUTCOMES:
Incidence rate of grade 2 or higher acute esophagitis | 3 months
  Assessed according to RTOG toxicity criteria.
Incidence rate of grade 3 or higher acute esophagitis assessed according to NCI-CTCAE v5.0 criteria | 3 months
  Assessed according to NCI-CTCAE v5.0 criteria
Incidence rate of grade 3 or higher acute esophagitis assessed according to RTOG toxicity criteria | 3 months
  Assessed according to RTOG toxicity criteria
Nutritional Assessment according to the Patient-Generated Subjective Global Assessment（PG-SGA） | 3 months
  PG-SGA scores range from 0 to 35, with higher scores indicating a greater risk of severe malnutrition.
Body weight | 3 months
Nutritional Risk | 3 months
  Assessed according to Nutritional Risk Screening 2002 (NRS 2002)
The duration period of esophagitis | 3 months
  The number of days of grade 2 or higher esophagitis
Opioid use | 3 months
  Measured by documented opioid use
Quality of life assessed by EORTC QLQ-C30 | 3 months
  EORTC QLQ-C30 scores range from 0 to 100, with higher scores indicating a better quality of life.
Quality of life assessed by FACT-L | 3 months
  FACT-L scores range from 0 to 108, with higher scores indicating a better quality of life.
Quality of life assessed by FACT-E Eating and Swallowing Subscales | 3 months
  FACT-E Eating and Swallowing Subscales scores range from 0 to 68, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Huai Liu, M.D., Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
Hospital policy